CLINICAL TRIAL: NCT07074444
Title: Albendazole, Tribendimidine, and Praziquantel for Clonorchiasis in Guangxi: A Randomized Controlled Trial Comparing Efficacy and Safety
Brief Title: Treatment of Clonorchiasis in Guangxi With Albendazole, Tribendimidine, and Praziquantel
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: People's Hospital of Guangxi Zhuang Autonomous Region (Other); Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-K0110
Record Dates: First submitted 2025-04-30; First posted 2025-07-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Clonorchiasis
Keywords: Clonorchiasis; Albendazole; Praziquantel; Egg clearance rate; tribendimidine
MeSH Terms: conditions — Clonorchiasis | interventions — Albendazole; tribendimidine; Praziquantel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Praziquantel (Active Comparator): Praziquantel tablets: Administer orally at 25 mg/kg per dose, three times daily (TID) for 2 consecutive days. The dose will be adjusted based on the participant's body weight. If the calculated dose results in a non-integer number of tablets, the dose will be adjusted to the nearest whole tablet according to the physician's recommendation.
  Interventions: Drug: praziquantel
- Albendazole (Experimental): Albendazole tablets: Administer orally at 10 mg/kg/day for 7 consecutive days. The daily dose will be administered in two divided doses. The dose will be adjusted based on the participant's body weight. If the calculated dose results in a non-integer number of tablets, the actual dose may be adjusted to the nearest whole tablet. The specific dose will be adjusted according to the physician's recommendation.
  Interventions: Drug: Albendazole
- Tribendimidine (Experimental): Tribendimidine enteric-coated tablets: Administer orally at 0.4 g once daily (QD) for 3 consecutive days.
  Interventions: Drug: Tribendimidine

INTERVENTIONS:
Drug: Albendazole — Participants receive albendazole tablets orally at a total daily dose of 10 mg/kg for 7 consecutive days. The daily dose will be administered in two divided doses. If the calculated dose results in a non-integer number of tablets, the dose will be adjusted to the nearest whole tablet as per the physician's recommendation.
  Arms: Albendazole
Drug: Tribendimidine — Patients receive tribendimidine enteric-coated tablets orally at 0.4 g once daily (QD) for 3 consecutive days.
  Arms: Tribendimidine
Drug: praziquantel — Participants receive praziquantel tablets orally at 25 mg/kg per dose, three times daily (TID) for 2 consecutive days. If the calculated dose results in a non-integer number of tablets, the dose will be adjusted to the nearest whole tablet as per the physician's recommendation.
  Arms: Praziquantel

SUMMARY:
The goal of this clinical trial is to evaluate and compare the efficacy and safety of three commonly used antiparasitic drugs-albendazole, tribendimidine, and praziquantel-for the treatment of clonorchiasis, a liver fluke infection acquired by consuming raw or undercooked freshwater fish.

This study aims to answer the following primary questions:

How effective is each drug in achieving parasitological cure, as measured by clearance of Clonorchis sinensis eggs in stool? What types and frequencies of adverse events are associated with each treatment?

Participants in this randomized, open-label trial will:

Be randomly assigned to receive one of the three study drugs according to a predefined dosing regimen.

Provide stool samples before treatment and at follow-up to assess for Clonorchis sinensis eggs.

Undergo a second round of the same treatment regimen and repeated stool examination if eggs are still detected after the first course.

Attend follow-up visits, which include symptom assessment, blood tests (hematology and liver function), and abdominal ultrasonography focusing on hepatobiliary changes.

Report any side effects, discomfort, or adverse reactions experienced during or after treatment.

The findings from this study will help inform optimal therapeutic strategies for clonorchiasis in outpatient clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years.
2. Confirmed diagnosis of Clonorchis sinensis infection based on the latest Expert Consensus on Diagnosis and Treatment of Food-Borne Parasitic Diseases (2023): detection of eggs or adult worms in stool or bile drainage fluid.
3. Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Known hypersensitivity or allergy to albendazole, praziquantel, or tribendimidine.
2. Electrocardiogram (ECG)-confirmed supraventricular tachycardia or atrial fibrillation.
3. Clinically or radiologically diagnosed neurocysticercosis (brain or spinal cord) or ocular cysticercosis (eye or orbit).
4. Presence of gallbladder stones or biliary tract obstruction as confirmed by abdominal ultrasound.
5. Individuals with severe hepatic, renal, or cardiac dysfunction, or with active peptic ulcer disease.
6. Pregnant or breastfeeding individuals, or those of reproductive potential (male or female) who are unwilling to use effective contraception during the study period and for 3 months following the last dose of study medication.
7. Anticipated loss to follow-up due to relocation, withdrawal of consent, or other factors affecting adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Egg Clearance Rate | From Day 30 to Day 60 after the last dose of treatment
  The primary outcome is the proportion of participants who test negative for Clonorchis sinensis eggs in all three stool samples collected at different time points post-treatment.

SECONDARY OUTCOMES:
Symptom Improvement Rate | Baseline and Day 31 (±1 day) after the last dose of treatment
  Symptom improvement will be assessed using a standardized symptom questionnaire or physician-recorded clinical evaluation. Typical symptoms associated with clonorchiasis-such as right upper abdominal pain, fatigue, and diarrhea-will be documented at baseline and again during the first follow-up visit, which takes place between Day 30 and Day 33 after the last dose of treatment. A symptom is considered improved if it shows significant relief or has completely resolved by that follow-up visit.
Hepatobiliary Ultrasonographic Improvement | Baseline and Day 31 (±1 day) after the last dose of treatment
  Among participants who show abnormal hepatobiliary findings on baseline abdominal ultrasonography (e.g., bile duct dilation, gallbladder wall thickening, or liver echogenicity changes), a repeat ultrasound will be performed at the follow-up visit (Day 30-33 after the last dose of treatment) to assess for resolution or improvement. Improvement is defined as partial or complete normalization of previously abnormal imaging features, as interpreted by a qualified radiologist.
Adverse Events (AEs) | From first dose to Day 30 (±1day) after the last dose of treatment
  Adverse events (AEs) will be collected from the initiation of treatment until the first follow-up visit, which occurs between Day 30 and Day 33 after the last dose of treatment. All events will be graded according to CTCAE version 5.0, and causality will be assessed using a five-level scale (definitely, probably, possibly, possibly not, and definitely not related). Serious adverse events (SAEs) will be documented and reported separately.
Proportion of Abnormal Hematology and Liver Function Results | Baseline and Day 31(±1 day) after the last dose of treatment
  Venous blood samples will be collected at baseline and follow-up (Day 30-33 after the last dose of treatment) for hematology and liver function tests. An abnormal result is defined as any value exceeding the laboratory reference range or deemed clinically significant by the investigator.
Drug Intolerance Rate | From first dose to Day 31 (+1 day) after the last dose of treatment
  Drug intolerance is defined as the inability to complete the planned treatment regimen due to serious adverse reactions, interruption of medication, or participant refusal. Data will be collected via participant self-report and investigator inquiry at the follow-up visit.

OTHER OUTCOMES:
Egg Clearance Rate After Second Treatment | From Day 30 to Day 60 after the last dose of second treatment]
  Among participants who remain egg-positive after the first treatment, a second course of the same antiparasitic regimen will be administered. Stool examinations will be performed on three separate days between Day 30 and Day 60 after the second treatment. Clearance is defined as negative egg detection in all three samples. The rate will be calculated among participants receiving the second treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hongliang Zhang, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (2):
- China (2):
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication, available upon request for 3 years.
Access Criteria: Researchers can gain access to the individual participant data (IPD) and supporting information by submitting a data sharing request proposal. The proposal must include a description of the planned analyses, including the statistical methods to be used. Proposals will be reviewed by an independent data access committee to ensure that the analyses are aligned with the study's objectives and meet ethical and scientific standards.
  To gain access, researchers must sign a data sharing agreement, which outlines the terms of use, including the intended use of the data, and any conditions for publication of results. Data sharing requests will be reviewed on a rolling basis, and researchers will be notified of the decision within 60 days of submission.